CLINICAL TRIAL: NCT03097016
Title: A Phase 1, Open-label, Single-dose Study to Assess the Pharmacokinetics (PK) of CC-122 in Subjects With Mild, Moderate and Severe Renal Impairment
Brief Title: A Study to Assess the Pharmacokinetics of CC-122 in Subjects With Mild, Moderate, and Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-122-CP-005
Record Dates: First submitted 2017-03-24; First posted 2017-03-31 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Renal Insufficiency
Keywords: Renal Impairment; Pharmacokinetics; CC-122; Mild; Moderate; Severe
MeSH Terms: conditions — Renal Insufficiency; Lymphoma, Follicular | interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single oral dose of 3 mg CC-122 (Experimental): All subjects will receive one 3 mg CC-122 capsule the morning of Day 1 which will be administered in the fasted state.
  Interventions: Drug: CC-122

INTERVENTIONS:
Drug: CC-122 — All subjects will receive one 3 mg CC-122 capsule the morning of Day 1 which will be administered in the fasted state.

SUMMARY:
Multi-center, open-label, single-dose study to assess the PK of a single oral dose of 3 mg CC-122 in subjects with mild, moderate, and severe renal impairment as compared to sex, age (± 15 years), and weight (± 20%) matched control subjects with normal renal function.

DETAILED DESCRIPTION:
This will be a multi-center, open-label, single-dose study to assess the PK of a single oral dose of 3 mg CC-122 in subjects with mild, moderate, and severe renal impairment as compared to sex, age (± 15 years), and weight (± 20%) matched control subjects with normal renal function. Estimated renal function for the purpose of group assignment will be determined at screening. Matched control subjects will have normal renal function, defined using the Cockcroft-Gault (C G) equation, as an estimated creatinine clearance (CLcr) of ≥ 90 mL/min. Subjects with impaired renal function will be classified by stage of renal impairment (mild, moderate, or severe) using estimated glomerular filtration rate (eGFR), calculated by the Modification of Diet in Renal Disease (MDRD) equation. Each group will enroll at least 2 subjects of each sex

During the course of the study, each subject will participate in a Screening period (Days - 21 to -2), Treatment Period (including baseline visit), and a follow-up telephone call between Days 11 to 18. Subjects will be screened for eligibility. Eligible subjects will return to the clinical site on Day 1 for baseline assessments, and will be domiciled at the clinical site from Day 1 to Day 4. PK samples will be collected through 72 hours post dose. Safety will be monitored throughout study.

The study will be conducted in compliance with the International Council on Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must satisfy all of the following criteria to be enrolled in the study:
* Subject must understand and voluntarily sign an Informed Consent Form prior to any study-related assessments/procedures being conducted.
* Subject is able to communicate with the Investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules and other protocol requirements.
* Subject is ≥ 18 and ≤ 80 years of age at the time of signing the informed consent.
* Subject has a body mass index between 18 and 40 kg/m2 (inclusive).
* Subject is afebrile
* Subject has a normal or clinically acceptable 12-lead Electrocardiogram at screening. In addition:

  * If male, subject has a QTcF value ≤ 470 msec at screening.
  * If female, subject has a QTcF value ≤ 480 msec at screening.
* Subject agrees to comply and abide by the requirements and restrictions outlined in the CC-122 Pregnancy Prevention Plan for Subjects in Clinical Trials.
* Female subjects must have been surgically sterilized (hysterectomy, bilateral oophorectomy, proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle-stimulating hormone level of> 40 IU/L at screening).
* Male subject must practice true abstinence* (which must be reviewed on a monthly basis, as applicable) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions (if applicable) and for at least 90 days following study drug discontinuation, even if he has undergone a successful vasectomy.

  * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Period abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Inclusion Criteria for Subjects with Mild, Moderate, or Severe Renal Impairment.

* Each subject with mild, moderate, or severe renal impairment must also meet ALL of the criteria listed below for entry:
* Subject has mild, moderate, or severe (not requiring dialysis) renal impairment as defined by Estimated glomerular filtration rate (eGFR) at screening.
* Subject has supine systolic BP: 90 to 180 mmHg, supine diastolic BP: 60 to 110 mmHg, and pulse rate: 40 to 110 bpm.
* Must be medically stable for at least 1 month before study drug administration with clinically acceptable medical history, Physical exam (PE), clinical laboratory tests, vital signs, and 12-lead ECGs consistent with the underlying stable mild moderate or severe renal impairment condition, as judged by the Investigator.
* Must be stable in concomitant medication regimen (defined as not starting a new medication[s] or a change in the dosage or frequency of the concomitant medication[s] within 7 days or 5 half-lives [whichever is longer] before dosing with study drug).

Inclusion Criteria for a Matched Healthy Subject

* Each matched healthy subject must meet ALL the criteria listed below for entry:
* Subject has supine systolic BP: 90 to 160 mmHg, supine diastolic BP: 50 to 100 mmHg, and pulse rate: 40 to 100 bpm
* Must be free of any clinically significant disease that would interfere with the study evaluations.
* Must have normal renal function, as defined by an eGFR ≥ 90 mL/min/1.73 m2 (calculated using the Modification of Diet in Renal Disease (MDRD) equation).
* Must match subjects in Group 1, 3, and 5 with respect to sex, age (± 15 years), and weight (± 20%).
* Must be in good health as determined by past medical history, PE, vital signs, ECG, and clinical laboratory safety tests. Clinical laboratory safety tests (i.e., hematology, chemistry, and urinalysis) and 12-lead ECGs must be within normal limits or clinically acceptable as judged by the Investigator.

Exclusion Criteria:

Exclusion Criteria for all subjects.

* The presence of any of the following will exclude a subject from enrollment:
* Subject has any condition or circumstance that prevents the subject from understanding and signing the Informed Consent Form.
* Subject has any condition that places the subject at an unacceptable risk from participating in the study or would confound the ability to interpret data from the study.
* Subject has any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, excretion, eg, bariatric procedure. Subjects with cholecystectomy and appendectomy may be included.
* Subject is a female of childbearing potential, pregnant, or breastfeeding.
* Subject donated blood or plasma within 8 weeks before dose administration to a blood bank or blood donation center.
* Subject has a history of alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 6 months before the first dose administration, or positive alcohol screen.
* Subject has a history of drug abuse (as defined by the current version of the DSM) within 6 months before the first dose administration, or positive drug screen that is not consistent with the patient's prescribed medication and or/medical history.
* Subject is known to have serum hepatitis or known to be a carrier of the hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV Ab) or have a positive result to the test for Human immunodeficiency virus (HIV) antibodies at screening. If a positive result for HCV AB is reported, the Investigator may assess the suitability of the subject based upon normal liver function test results and either no history of Hepatitis C, or documented sustained viral response (ie, undetectable HCV viral load during and 12 weeks after completion of accepted HCV treatment). If the subject meets both criteria, and the Investigator determines this as acceptable, the subject can be considered for enrollment into the trial.
* Subject was exposed to an investigational drug (new chemical entity) within 30 days before dosing, or 5 half-lives of that investigational drug, if known (whichever is longer).
* Subject smokes more than 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
* Subject has a history of multiple drug allergies or drug-related anaphylaxis.
* Subject used approved medications or herbal medicines that are moderate or strong cytochrome P450 (CYP)1A2 or 3A4/5 inducers and/or inhibitors (including St. John's wort) within 14 days or 5 half-lives of dosing, whichever is longer. The Indiana University "Cytochrome P450 Drug Interaction Table" should be utilized to determine inhibitors and/or inducers of CYP1A2 and CYP3A4/5. (http://medicine.iupui.edu/clinpharm/ddis/table.aspx).
* Subject has received vaccination (excluding seasonal flu vaccination) within 90 days of dosing.
* Subject is part of the staff personnel or a family member of the investigational study staff.

Exclusion Criteria for Subjects with Mild, Moderate, or Severe Renal Impairment.

* Each renal impairment subject will be excluded from entry if ANY of the criteria listed below are met:
* Any serious and or unstable medical condition occurring within 3 months prior to signing the Informed Consent Form (excluding stable renal impairment and associated comorbidities).
* Any clinically significant laboratory abnormality not related to renal impairment and related complications.
* History of renal transplant.
* Subjects with renal impairment should be excluded from study if laboratory values are outside the following ranges and, in the opinion of the Investigator, are considered to prevent the subject from safely completing the study:

Exclusion Criteria for Subjects with Mild, Moderate, or Severe Renal Impairment.

* Each matched healthy subject will be excluded from entry if ANY of the criteria listed below are met:
* Subject has any clinically significant laboratory abnormality that in the opinion of the Investigator, is considered to prevent the subject from safely completing the study.
* Subject has any unstable clinically significant illness within 3 months prior to the study.
* Subject used any prescribed systemic or topical medication within 30 days prior to signing of the Informed Consent Form.
* Subject used any non-prescribed systemic or topical medication within 7 days prior to signing of the Informed Consent Form (with the exception of vitamin/mineral supplements).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2017-12-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Tmax | up to 72 hours
  Time to Observed maximum serum concentration (Cmax)
Pharmacokinetics - Cmax | up to 72 hours
  Observed maximum serum concentration (Cmax)
Pharmacokinetics - AUC0-t | up to 72 hours
  Area under the serum concentration-time curve calculated from time zero to the last measured time point
Pharmacokinetics - AUC0-∞ | up to 72 hours
  Area under the serum concentration-time curve calculated from time zero to infinity
Pharmacokinetics - t1/2 | Up to 72 hours
  Terminal elimination half-life
Pharmacokinetics - CL/F | Up to 72 hours
  Apparent clearance of drug from serum when dosed orally
Pharmacokinetics - Vz/F | Up to 72 hours
  Apparent volume of distribution when dosed subcutaneously during the terminal phase
Pharmacokinetics - CLR | Up to 72 hours
  Renal Clearance
Pharmacokinetics - Ae | Up to 72 hours
  Amount of excretion

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to 40 days
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopoulos, MD, Study Director — Celgene
Locations (2):
- United States (2):
  - DaVita Clinical Research, Lakewood, Colorado
  - DaVita Clinical Research, Minneapolis, Minnesota